CLINICAL TRIAL: NCT01877993
Title: The Association of Acetylcholine-induced Coronary Artery Spasm With the Blood Pressure Level
Brief Title: The Effect of Autonomic Function on Coronary Vasomotion
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Collaborators: Korea Institute of Science and Technology (Other)
Responsible Party: Principal Investigator, Hong Seog Seo, Professor of Medicine, Korea University
Other Study IDs: BP-CAS
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Coronary Artery Spasm; Autonomic Dysfunction
Keywords: coronary artery spasm; pathophysiology; atrioventricular block; blood pressure; autonomic nervous function
MeSH Terms: conditions — Coronary Vasospasm; Primary Dysautonomias; Atrioventricular Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Autonomic nerve function is involved in both blood pressure (BP) regulation and the pathogenesis of coronary artery spasm (CAS), but few studies have been published about the relationship between CAS and BP, with the exception of studies that explore hypertension as a risk factor for CAS. The purpose of this study was to investigate the incidence of CAS and atrioventricular (AV) block in association with BP level. The investigators will register consecutive patients who underwent coronary angiography with an acetylcholine (Ach)-induced provocation test from November 2004 to May 2012. The investigators exclude from the patients who were taking antihypertensive drugs or who had a documented history of cardiovascular disease in order to avoid the confounding effects of cardiovascular medications on coronary vasomotion. CAS is defined as >70% luminal narrowing on Ach provocation and /or concurrent chest pain. The study population will be divided into quartiles of rising systolic BP and diastolic BP. The incidence of Ach-induced CAS according to each systolic BP/diastolic BP quartile will be evaluated.

DETAILED DESCRIPTION:
A total of consecutive patients in the CAS registry of the Cardiovascular Center at Korea University Guro Hospital and who had resting chest pain without significant coronary lesions (luminal narrowing <50%) underwent a provocation test with Ach infusion during coronary angiography from November 2004 to May 2012 will be registerd. Among them, patients with documented cardiovascular disease and/or any other serious medical condition, such as an increased serum creatinine level (>2mg/dl), will be excluded. Patients will be excluded due to incomplete data. The study population will be divided into quartiles based on rising systolic BP, diastolic BP, and pulse pressure. Each group will be defined as following criteria: 1) group 1: systolic BP <117mmHg, diastolic BP <69mmHg, and pulse pressure <42mmHg; 2) group 2: systolic BP 117-130 mmHg, diastolic BP 69-77 mmHg, and pulse pressure 42-51mmHg; 3) group 3: systolic BP 131-141 mmHg, diastolic BP 78-86 mmHg, and pulse pressure 52-61mmHg; and 4) group 4: systolic BP >141 mmHg, diastolic BP >86 mmHg, and pulse pressure >61mmHg. CAS+Chest Pain means>70% luminal narrowing on Ach provocation test. and/or concurrent typical chest pain. BP was measured with a noninvasive BP monitoring device with the patient lying on the angiographic table after a five-minute rest (Patient monitoring system, NP 30:Philips, Amsterdam, The Netherlands). The first reading was discarded, and the mean of the next two consecutive readings was used. Next, coronary angiography was performed. Hypertension is defined as systolic BP ≥140mmHg and/or diastolic BP ≥90mmHg on at least two consecutive readings in the outpatient clinic. Patients taking antihypertensive medications are also categorized as hypertensives. Other Risk factors for CAS examined in this study include hyperlipidemia (total cholesterol level ≥200mg /dl or current medication with lipid-lowering drugs), diabetes (fasting blood glucose≥126mg /dl, and/or glycated Hemoglobin A1c level more than 6.5% or current use of medications), current smoker (active smoking within the past 12 months), and current alcohol user (at least 1 alcohol drinking a week).

ELIGIBILITY:
Inclusion Criteria:

* patients had resting chest pain without significant coronary lesions (luminal narrowing <50%) underwent a provocation test with Ach infusion during coronary angiography.

Exclusion Criteria:

* patients with documented cardiovascular disease and/or any other serious medical condition, such as an increased serum creatinine level (>2mg/dl), patients with incomplete data, and patients who had been diagnosed with hypertension or were currently using antihypertensive medications.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 5,304 consecutive patients in the CAS registry of the Cardiovascular Center at Korea University Guro Hospital
Sampling Method: Non-Probability Sample
Enrollment: 2169 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
development of significant CAS | during the Ach provocation test
  During the Ach provocation test, significant CAS was recorded when present, and we recorded whether it was associated with any of the four following criteria: 1) chest pain only during Ach provocation test 2) >70% luminal narrowing on coronary angiography and concurrent typical chest pain;3) >70% luminal narrowing on coronary angiography and/or concurrent chest pain and EKG changes(ST-segment elevation or depression ≥1mm); 4) >90% luminal narrowing induced by A3 dose on coronary angiography and/or concurrent chest pain.

SECONDARY OUTCOMES:
Transient high-grade AV block | occurred in response to Ach injection
  Transient high-grade AV block that occurred in response to Ach injection is defined as such if it consisted of multiple sequential P waves that should conduct, but did not.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Seog Seo, MD, Ph., Principal Investigator — Korea University Guro Hospital
Locations (3):
- South Korea (3):
  - Department of Internal Medicine, Division of Cardiology, Sanbon Hospital, Wonkwang University, Gunpo, Gyeonggi-do
  - Hong Seog Seo, Seoul
  - Korea Institute of Science and Technology, Seoul